CLINICAL TRIAL: NCT01580579
Title: Clinical, Biochemical, Dosimetric and Functional Respiratory Predictors of Radiation Pneumonitis in Locally Advanced Lung Cancer (Stages IIIa and IIIb) Treated With Chemotherapy and Radiotherapy
Brief Title: Predictors of Radiation Pneumonitis in Locally Advanced Lung Cancer Treated With Chemoradiation
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, Chief of Thoracic Oncology Department, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: INCANOGAR2012-JA2
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Radiation; Adverse Effect, Pneumonitis
Keywords: Radiation pneumonitis; locally advanced lung cancer; Respiratory function tests
MeSH Terms: conditions — Pneumonia; Radiation Pneumonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- locally advanced lung cancer: Patients with locally advanced lung cancer who are candidates to chemoradiation

SUMMARY:
Lung cancer [LC] is the leading cause of cancer death worldwide. The standard treatment of locally advanced lung cancer unresectable or marginally resectable is combination therapy with radical or preoperative chemoradiation. The local control rates and survival with this treatment modality have increased by more than 30%. Radiotherapy [RT] with technical molded 3D [3D-CRT, Three-Dimensional Conformal Radiation Therapy] or IMRT [intensity-modulated radiation therapy] has allowed that the total dose of radiation has increased which leads to a direct benefit on the results treatment.

Between 17-30% of patients are susceptible to pneumonitis due to radiation [NR]. This complication may appear at the end of the RT or up to 6 months after the treatment. In severe cases, mortality can reach 50%.

It's well known that in various diseases, functional abnormalities precede the clinical manifestations. The degree of pulmonary failure secondary to RT is measured following the standards of the Radiation Therapy Oncology Group who ranks in degrees [0 to 4].

Not precisely known factors that influence the development of NR.

DETAILED DESCRIPTION:
Objectives:

To evaluate the effect of chemotherapy and thoracic radiotherapy on pulmonary function and identify predictors of radiation pneumonitis in locally advanced lung cancer [stages IIIA and IIIB].

Hypothesis:

Respiratory function tests may predict the development of radiation pneumonitis in patients with locally advanced lung cancer who receive radical treatment with chemoradiation.

Methods Prospective cohort study with patients with locally advanced lung cancer of the Lung Cancer Clinic of the National Cancer Institute [INCAN]. Patients will receive weekly paclitaxel 50 mg and carboplatin AUC 2 with concomitant radiotherapy 44-63 Gy (22-33 fractions). Followup of lung function tests at baseline, during treatment with radiotherapy and will be carried out on 4 more occasions.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must have understood and signed informed consent
* Histopathological diagnosis of locally advanced lung cancer [IIIA-cT2N1-2, cT3N1-2, cT4N0, M0o IIIB: cT2N3, cT3N3, cT4N1-3, M0]. They may also include patients with oligometastatic disease[M1] candidates for chemoradiation
* Any histology
* Medical tests: white blood cell count ≥ plasma 3,000 / mm3, platelets ≥ 100,000 / mm 3, hemoglobin ≥ 12 g / dl, serum creatinine ≤ 1.5 mg / dl, total bilirubin ≤ 1.5, transaminases [ ≤ 2.5 times the upper limit of normal [ULN], alkaline phosphatase <5 ULN.
* Age ≥ 18 years.
* General condition score according to ECOG 0 to 2 or a ≥ 60% Karnofsky.
* Estimated life expectancy with treatment of at least 24 weeks.

Exclusion criteria:

* Uncontrolled concurrent diseases.
* History of previous radiotherapy to the primary site.
* Pregnant or breast-feeding.
* Use of anticoagulants in therapeutic doses
* Intercurrent Malignancies, except dormant basal cell carcinoma in skin, carcinoma in situ of the cervix
* Invasive cancer unless the background was at least 5 years and the disease-free status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced lung cancer candidates to receive treatment with chemoradiation that will receive treatment in the National Cancer Institute in Mexico City.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evaluate pulmonary function after chemoradiation treatment in locally advanced NSCLC patients. | January 2012 to December 2014

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — Instituto de Cancerología
Locations (1):
- Instituto Nacional de Cancerología de México, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kim M, Lee J, Ha B, Lee R, Lee KJ, Suh HS. Factors predicting radiation pneumonitis in locally advanced non-small cell lung cancer. Radiat Oncol J. 2011 Sep;29(3):181-90. doi: 10.3857/roj.2011.29.3.181. Epub 2011 Sep 30. PMID 22984669
- [Background] Noble PW, Barkauskas CE, Jiang D. Pulmonary fibrosis: patterns and perpetrators. J Clin Invest. 2012 Aug;122(8):2756-62. doi: 10.1172/JCI60323. Epub 2012 Aug 1. PMID 22850886
- [Background] Kong FM, Hayman JA, Griffith KA, Kalemkerian GP, Arenberg D, Lyons S, Turrisi A, Lichter A, Fraass B, Eisbruch A, Lawrence TS, Ten Haken RK. Final toxicity results of a radiation-dose escalation study in patients with non-small-cell lung cancer (NSCLC): predictors for radiation pneumonitis and fibrosis. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1075-86. doi: 10.1016/j.ijrobp.2006.01.051. Epub 2006 May 2. PMID 16647222
- [Derived] Torre-Bouscoulet L, Arroyo-Hernandez M, Martinez-Briseno D, Munoz-Montano WR, Gochicoa-Rangel L, Bacon-Fonseca L, Perez-Padilla R, Vergara E, Garcia-Sancho C, Lozano-Ruiz F, Fernandez-Plata R, Guzman-Barragan A, Arrieta O. Longitudinal Evaluation of Lung Function in Patients With Advanced Non-Small Cell Lung Cancer Treated With Concurrent Chemoradiation Therapy. Int J Radiat Oncol Biol Phys. 2018 Jul 15;101(4):910-918. doi: 10.1016/j.ijrobp.2018.04.014. Epub 2018 Apr 12. PMID 29976503
- [Derived] Torre-Bouscoulet L, Munoz-Montano WR, Martinez-Briseno D, Lozano-Ruiz FJ, Fernandez-Plata R, Beck-Magana JA, Garcia-Sancho C, Guzman-Barragan A, Vergara E, Blake-Cerda M, Gochicoa-Rangel L, Maldonado F, Arroyo-Hernandez M, Arrieta O. Abnormal pulmonary function tests predict the development of radiation-induced pneumonitis in advanced non-small cell lung Cancer. Respir Res. 2018 Apr 24;19(1):72. doi: 10.1186/s12931-018-0775-2. PMID 29690880